CLINICAL TRIAL: NCT07159217
Title: A Prospective Exploratory Phase II Study of Disitamab Vedotin Plus Lenvatinib and PD-1 Inhibitors for the Treatment of HER2-positive Advanced Biliary Tract Cancer
Brief Title: Disitamab Vedotin Plus Lenvatinib and PD-1 Inhibitors for Treating HER2-positive Advanced Biliary Tract Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: K8721
Record Dates: First submitted 2025-08-18; First posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Biliary Tract Cancer; Disitamab Vedotin; Lenvatinib; Immune Checkpoint Inhibitors
Keywords: Biliary tract cancer; Disitamab vedotin; Lenvatinib; Immune checkpoint inhibitors
MeSH Terms: conditions — Biliary Tract Neoplasms | interventions — disitamab vedotin; lenvatinib; pembrolizumab; toripalimab; camrelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Disitamab vedotin combined with lenvatinib and PD-1 inhibitor (Experimental): Disitamab vedotin combined with lenvatinib and PD-1 inhibitor (Pembrolizumab or Toripalimab or Camrelizumab)
  Interventions: Drug: Disitamab Vedotin; Drug: Lenvatinib; Drug: Pembrolizumab; Drug: Toripalimab; Drug: Camrelizumab

INTERVENTIONS:
Drug: Disitamab Vedotin — 2.0 mg/kg administered intravenously every three weeks
Drug: Lenvatinib — ≥60 kg: 12 mg once daily, or <60 kg: 8 mg once daily
Drug: Pembrolizumab — 200 mg intravenously every three weeks
Drug: Toripalimab — 240 mg intravenously every three weeks
Drug: Camrelizumab — 200 mg intravenously every three weeks

SUMMARY:
This trial is a single-arm exploratory phase II clinical study initiated by the investigator.

Subjects who met the research criteria were screened and enrolled to receive the treatment regimen of disitamab vedotin combined with lenvatinib and PD-1 inhibitor. During the treatment process, the researchers closely followed up, strictly evaluated the efficacy, assessed the efficacy and safety of the subjects after receiving the combined treatment, evaluated the subjects until progression occurred, and observed their objective response rate, progression-free survival, overall survival, disease control rate, duration of response, and safety evaluation.

ELIGIBILITY:
Inclusion criteria:

1. Participants who voluntarily participate in this study, sign the written informed consent, and are able to comply with the protocol.
2. Age ≥ 18 years and any gender.
3. Histologically or cytologically confirmed unresectable locally advanced or metastatic biliary tract cancer (BTC), including intrahepatic cholangiocarcinoma (ICC), extrahepatic cholangiocarcinoma (ECC), and gallbladder cancer (GBC).
4. At least one measurable lesion (according to RECIST 1.1).
5. ECOG performance status score of 0-1.
6. Child-Pugh score ≤ 7 .
7. HER2 expression confirmed by: Immunohistochemistry (IHC 2+ or 3+); or Fluorescence in situ hybridization (FISH) with HER2/CEP17 ratio ≥2.0; or Next-generation sequencing (NGS) showing HER2 amplification.
8. No prior HER2-targeted therapy (including antibody-based agents, small-molecule TKIs, or antibody-drug conjugates) before randomization.
9. Expected survival > 12 weeks.
10. Adequate hematological and major organ function.

Exclusion criteria：

1. Histological or cytological diagnosis of combined hepatocellular-cholangiocarcinoma (cHCC-CCA), mucinous adenocarcinoma, sarcoma, or neuroendocrine tumors.
2. Pregnant women (positive pregnancy test before medication) or lactating women.
3. Known allergy or intolerance to disitamab vedotin, lenvatinib, PD-1 inhibitors, or their excipients.
4. History of other active malignancies within 5 years prior to screening.
5. Presence of central nervous system metastasis and/or leptomeningeal metastasis.
6. Unhealed severe wounds, active ulcers, or untreated fractures.
7. Administration of live vaccines within 30 days prior to randomization.
8. Active autoimmune disease or history of autoimmune disease.
9. Presence of clinically significant gastrointestinal disorders.
10. Presence of clinically significant cardiovascular or cerebrovascular diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2025-08-30 (Estimated); Primary Completion 2027-05-31 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
ORR, objective response rate | 12 months after the last subject is enrolled

SECONDARY OUTCOMES:
PFS, progression free survival | 12 months after the last subject is enrolled
OS, overall survival | 12 months after the last subject is enrolled
DCR, disease control rate | 12 months after the last subject is enrolled
DoR, duration of response | 12 months after the last subject is enrolled
Adverse events (AE) and serious adverse events (SAE) | 12 months after the last subject is enrolled
  To evaluate safety, incidence and outcome of adverse events (AE), and serious adverse events (SAE)

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese Academy of Medical Sciences, Peking Union Medical College Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shi F, Liu Y, Zhou X, Shen P, Xue R, Zhang M. Disitamab vedotin: a novel antibody-drug conjugates for cancer therapy. Drug Deliv. 2022 Dec;29(1):1335-1344. doi: 10.1080/10717544.2022.2069883. PMID 35506447